CLINICAL TRIAL: NCT01348347
Title: An Open-label Phase I Study of Once Every Three Weeks Intravenous Treatment With BI 6727 in Japanese Patients With Advanced Solid Tumours
Brief Title: BI 6727 (Volasertib) Monotherapy Phase I Trial in Japanese Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230.15
Record Dates: First submitted 2011-04-29; First posted 2011-05-05 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BI 6727

ARMS (1):
- Volasertib (Experimental): Patient to receive low, middle and high doses of Volasertib IV
  Interventions: Drug: Volasertib, low dose, d1q3w; Drug: Volasertib, middle dose, d1q3w; Drug: Volasertib, high dose, d1q3w

INTERVENTIONS:
Drug: Volasertib, low dose, d1q3w — Patient to receive low dose of Volasertib IV
Drug: Volasertib, middle dose, d1q3w — Patient to receive middle dose of Volasertib IV
Drug: Volasertib, high dose, d1q3w — Patient to receive high dose of Volasertib IV

SUMMARY:
This open-label phase I dose escalation trial, 1230.15, is the first trial with Volasertib in Japanese advanced cancer patients. The trial will investigate the maximum tolerated dose (MTD), safety, tolerability, and preliminary efficacy of this specific polo-like kinase 1 (Plk1) inhibitor in advanced cancer patients.

ELIGIBILITY:
Inclusion criteria:

1. Patients with histologically or cytologically confirmed according to the discretion of the investigator
2. Patients who have advanced, non-resectable and/or metastatic solid tumours according to the discretion of the investigator
3. Patients who have failed conventional treatment, or for whom no therapy of proved efficacy exists, or who are not amenable to established forms of treatment according to the discretion of the investigator
4. Age >=20 years old at the time of informed consent
5. Written informed consent
6. Life expectancy of at least 12 weeks according to the discretion of the investigator
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
8. Recovery to Common Terminology Criteria for Adverse Events (CTCAE) grade =1 of therapy-related toxicities from previous chemo-, hormonal-, immuno-, or radiotherapy (except alopecia and hyperpigmentation)
9. Adequate bone marrow, renal and hepatic function;

   * Neutrophil count: more than 1500/mm3
   * Platelet count: more than 100 000/mm3
   * Haemoglobin: more than 9.0 g/dL
   * Total bilirubin: less than 1.5 times the upper limit of normal (ULN)
   * Aspartate amino transferase (AST): less than 2.5 × ULN
   * Alanine amino transferase (ALT): less than 2.5 × ULN
   * Serum creatinine: less than 1.5 × ULN
10. Patients who can be hospitalised during the first course

Exclusion criteria:

1. Major surgery within 4 weeks prior to registration or the side effects/toxicities of such surgery that have not recovered to CTCAE grade =1
2. Known seropositivity to human immunodeficiency virus (HIV) antibody, hepatitis B antigen or hepatitis C antibody
3. Accumulation of coelomic fluid (e.g. pleural effusion, ascites fluid) requiring treatment during the trial (Patients are eligible if treated curatively and with no evidence of recurrence.)
4. Current symptomatic brain metastases or patients who require treatment of the brain metastases
5. Previous double cancers. Other tumours (except for non-invasive and/or non-melanomatous skin cancer, completely removed in situ carcinoma of the epithelium or mucosa) treated curatively and with no evidence of recurrence for at least 5 years prior to the initial study treatment will be eligible.
6. Known history of cardiac dysfunction;

   * Correction of QT intervals according to Fridericias formula (QTc) over 470 ms
   * History of unstable angina pectoris within 6 months or current unstable angina pectoris
   * History of myocardial infarction within 6 months
   * Arrhythmia currently required active therapy
   * Previous and current cardiac failure
   * History of other clinically significant cardiac diseases according to the discretion of the investigator
7. Pregnant or breastfeeding women
8. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. implants, injectables, combined oral contraceptives, some intrauterine devices, vasectomised partner, or condoms) during the trial and for at least 6 months after the end of active therapy. Women who are sexually active are premenopausal female patients. Premenopausal female patient is defined as the patient who observed menses within 12 months except for an alternative medical cause. Women who underwent an operation for sterilisation is excluded for this criteria.
9. Treatment with other investigational drugs within the past 4 weeks before registration or concomitantly with this trial (except for present trial drug)
10. Chemo-, radio-, immuno-, or molecular-targeted therapy within the past 4 weeks before registration or concomitantly with this trial. This restriction does not apply to bisphosphonates.
11. Patients unable to comply with the protocol according to the discretion of the investigator or sub-investigators
12. Current alcohol abuse or drug abuse according to the discretion of the investigator
13. Patients who are inappropriate for this trial by the discretion of investigator or sub-investigators (e.g. uncontrolled diabetes mellitus, evidence of serious active infection, medically significant abnormal laboratory finding, etc.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04-25 (Actual); Primary Completion 2012-08-27 (Actual); Study Completion 2014-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1230.15.001 National Cancer Center Hospital,, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Derived] Nokihara H, Yamada Y, Fujiwara Y, Yamamoto N, Wakui H, Nakamichi S, Kitazono S, Inoue K, Harada A, Taube T, Takeuchi Y, Tamura T. Phase I trial of volasertib, a Polo-like kinase inhibitor, in Japanese patients with advanced solid tumors. Invest New Drugs. 2016 Feb;34(1):66-74. doi: 10.1007/s10637-015-0300-0. Epub 2015 Dec 2. PMID 26627079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 patients were treated and analysed.
Pre-assignment Details: This was an open-label, uncontrolled, dose escalation phase I study of once every three weeks intravenous treatment with BI 6727(volasertib) in Japanese patients with advanced solid tumours.
Groups:
- Volasertib 200 mg Cohort: Volasertib 200 mg was infused intravenously (over 2 hours) on Day 1 in a 3-week treatment course.
- Volasertib 300 mg Cohort: Volasertib 300 mg was infused intravenously (over 2 hours) on Day 1 in a 3-week treatment course.
- Volasertib 350 mg Cohort: Volasertib 350 mg was infused intravenously (over 2 hours) on Day 1 in a 3-week treatment course.
Period: Overall Study
Arm/Group | Volasertib 200 mg Cohort | Volasertib 300 mg Cohort | Volasertib 350 mg Cohort
Started | 3 | 6 | 6
Completed | 0 | 0 | 0
Not Completed | 3 | 6 | 6
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Progressive disease | 2 | 5 | 5

BASELINE CHARACTERISTICS:
Population: The treated set(TS) - All patients who received ≥1 dose of study medication (volasertib) were included in the treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Volasertib 200 mg Cohort | Volasertib 300 mg Cohort | Volasertib 350 mg Cohort | Total
Number analyzed (Participants) | 3 | 6 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (7.9) | 58.8 (11.4) | 60.8 (8.6) | 61.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 2 | 6 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in Process for the Determination of the Maximum Tolerated Dose (MTD).
Description: The following drug-related adverse events (AE) were defined as DLT;
  1. Haematological toxicities: CTCAE(Common Terminology Criteria for Adverse Events) grade 4 neutropenia persisted for 7 or more days, CTCAE grade 4 thrombocytopenia or CTCAE grade 3 thrombocytopenia requiring blood transfusion.
  2. Non-haematological toxicities: CTCAE grade ≥3 non-haematological toxicities. The following toxicity with neutropenia was defined as DLT.- CTCAE grade 3 febrile neutropenia persisted for over 2 days, Clinically significant laboratory abnormalities of CTCAE grade ≥3 persisted for over 3 days. The following laboratory abnormalities should be defined as DLT. - Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): >5.0 × ULN persisted for 7 days or longer - Creatinine: >3.0 × upper limit of normal(ULN) (if the creatinine abnormality was observed even once) - Persistent electrolyte abnormality assessed by the investigator.
Time Frame: 21 days
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Volasertib 200 mg Cohort | Volasertib 300 mg Cohort | Volasertib 350 mg Cohort
Number analyzed (Participants) | 3 | 6 | 6
Participants | 0 | 0 | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Volasertib
Description: Maximum tolerated dose (MTD) of volasertib was the highest dose tested at which DLT was developed in not more than 1 of 6 patients in the course 1.
Time Frame: 21 days
Population: as for baseline characteristics
Measure: Number; unit: mg
Groups:
- Volasertib Cohort: Volasertib with 200mg, 300mg and 350mg were infused intravenously (over 2 hours) on Day 1 in a 3-week treatment course .
Arm/Group | Volasertib Cohort
Number analyzed (Participants) | 15
mg | 300

3. Secondary Outcome: Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1
Description: Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1: Unconfirmed objective response. The patients with complete response (CR) or partial response (PR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by magnetic resonance imaging (MRI): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Volasertib 200 mg Cohort | Volasertib 300 mg Cohort | Volasertib 350 mg Cohort
Number analyzed (Participants) | 3 | 6 | 6
Participants
  No | 3 | 6 | 5
  Yes | 0 | 0 | 1

4. Secondary Outcome: Disease Control Rate According to RECIST v1.1
Description: Disease control rate according to RECIST v1.1 - Unconfirmed disease control. The patients with complete response (CR), partial response (PR) or stable disease (SD).
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Volasertib 200 mg Cohort | Volasertib 300 mg Cohort | Volasertib 350 mg Cohort
Number analyzed (Participants) | 3 | 6 | 6
Participants
  No | 0 | 1 | 2
  Yes | 3 | 5 | 4

5. Secondary Outcome: Cmax of Volasertib (BI 6727)
Description: Maximum concentration of an analyte in plasma
Time Frame: Pharmacokinetic (PK) plasma samples were taken at: 5 minutes predose, 1hour, 2hours (h), 3h, 4h, 8h, 24h, 48h, 72h, 96h, 168h and 336h of course1.
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Volasertib 200 mg Cohort | Volasertib 300 mg Cohort | Volasertib 350 mg Cohort
Number analyzed (Participants) | 3 | 6 | 6
ng/mL | 398 (17.6) | 501 (17.7) | 615 (37.7)

6. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity) of Volasertib (BI 6727)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity) of Volasertib (BI 6727).
Time Frame: PK plasma samples were taken at: 5 minutes predose, 1hour, 2hours (h), 3h, 4h, 8h, 24h, 48h, 72h, 96h, 168h and 336h of course1.
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Volasertib 200 mg Cohort | Volasertib 300 mg Cohort | Volasertib 350 mg Cohort
Number analyzed (Participants) | 3 | 6 | 6
ng*h/mL | 4350 (25.0) | 5300 (16.3) | 7260 (14.9)

7. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 up to the Last Quantifiable Data Point (AUC0-tz) of Volasertib (BI 6727)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 up to the last quantifiable data point (AUC0-tz) of Volasertib (BI 6727).
Time Frame: as for outcome 6
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Volasertib 200 mg Cohort | Volasertib 300 mg Cohort | Volasertib 350 mg Cohort
Number analyzed (Participants) | 3 | 6 | 6
ng*h/mL | 4000 (19.1) | 5100 (16.6) | 6900 (15.5)

ADVERSE EVENTS:
Time Frame: From the day of informed consent(-14 days) until the follow-up visit, 72 days.
Arm/Group | Volasertib 200 mg Cohort | Volasertib 300 mg Cohort | Volasertib 350 mg Cohort
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib 200 mg Cohort (N=3) | Volasertib 300 mg Cohort (N=6) | Volasertib 350 mg Cohort (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib 200 mg Cohort (N=3) | Volasertib 300 mg Cohort (N=6) | Volasertib 350 mg Cohort (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 5 | 6
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 6 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 2 | 4
Injection site reaction (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3
Blood albumin decreased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
250 mg dose of Volasertib was planned, as needed. However the 250 mg intermediate cohort had not been implemented in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.